CLINICAL TRIAL: NCT04225338
Title: Retrospective Study of Patients Undergoing Percutaneous Intervention of the Transplant Renal Artery Stenosis (TRAS Study)
Brief Title: Retrospective Study of Patients Undergoing Percutaneous Intervention of the Transplant Renal Artery Stenosis
Acronym: TRAS
Status: Completed | Type: Observational
Sponsor: Adriano Henrique Pereira Barbosa (Other)
Responsible Party: Sponsor-Investigator, Adriano Henrique Pereira Barbosa, Principal Investigator, Federal University of São Paulo
Organization: Federal University of São Paulo (Other)
Other Study IDs: FUSaoPaulo TRAS
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Transplant Renal Artery Stenosis
Keywords: renal transplantation; transplated renal artery stenosis; percutaneous intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Renal transplantation is the standard treatment for patients with end-stage chronic kidney disease because it is effective in reducing the morbidity and mortality. Despite of the satisfactory results, some patients evolve with graft dysfunction and refractory hypertension due to transplanted renal artery stenosis (TRAS). TRAS is the main vascular complication of patients undergoing kidney transplantation, with a reported incidence ranging 1 to 23% in the different series in the literature, depending on the definition and diagnostic techniques used, manifesting most commonly between the 3rd month and the 2nd year after transplantation.

Percutaneous intervention of TRAS is widely accepted as a viable treatment option, but there are few long-term data on patients undergoing angioplasty. The aim of this study was to evaluate long term outcomes clinical in patients with TRAS underwent to percutaneous intervention with or without stent.

DETAILED DESCRIPTION:
Renal transplantation is the standard treatment for patients with end-stage chronic kidney disease, as it is effective in reducing the morbidity and mortality of patients in this condition. Despite satisfactory results, some patients have graft dysfunction and difficult-to-control hypertension, with the main cause of transplanted renal artery stenosis (TRAS).

The incidence of TRAS varies from 1 to 23% in the various series in the literature, depending on the definition and diagnostic techniques used, most commonly occurring between the 3rd month and the 2nd year after transplantation. However, it may present at any time with refractory hypertension and / or graft dysfunction in the absence of rejection, ureteral obstruction or infection.

About 50% of TRAS cases occur at the anastomosis site and there seems to be no relationship with the type of anastomosis, whether end-to-end or end-to-side. TRAS is generally a consequence of clamp perfusion injury, incorrect suture technique, or fibrotic inflammatory reaction to suture material. Other factors attributed to TRAS are secondary to graft rejection, cytomegalovirus infection, and cadaveric donor graft. The last two factors are controversial in the literature. Late TRAS is related to progressive atherosclerosis.

The diagnosis of TRAS is made by clinical manifestations and / or by complementary exams. In addition to refractory hypertension, patients with TRAS may have increased serum creatinine, sudden graft deterioration and acute pulmonary edema. Color Doppler ultrasonography is the most commonly used method due to its easy access, low cost and does not require the use of contrast or radiolabels. However, its biggest limitation is the heavy reliance on operator expertise. It has a sensitivity of 87 to 94% and a specificity of 86 to 100%. TRAS is suspected when Doppler ultrasound has a peak systolic velocity (PSV) above 180 cm / s and a resistance index <0.50.

Computed tomography provides three-dimensional images that may be superior to those of selective angiography, with the advantage of not requiring arterial puncture and requiring less contrast. Nuclear magnetic resonance is even superior to tomography, with a sensitivity of 67 to 100% and specificity of 75 to 100%. However, its availability is still limited, besides presenting high costs.

Renal arteriography is the gold standard for the diagnosis of TRAS. However, there is a need for high contrast volumes, which can precipitate acute renal failure, particularly in patients who already have renal dysfunction. Three-dimensional rotational angiography (3D-RA) appears as an auxiliary tool that can minimize the deleterious effects of contrast. The measurements obtained by 3D-RA showed a strong correlation with the measurements made by conventional angiography, demonstrating equivalent accuracy, without the need for additional projections, helping to perform the intervention.

Complications arising from transplanted kidney arteriography are puncture site hematomas, pseudoaneurysms, thromboembolism, arteriovenous fistulas, iliac artery dissection, graft artery dissection, occurring in less than 10% of cases. Due to the substantial risks and high costs, arteriography cannot be considered a screening method and is only indicated when a stenosis is suspected based on noninvasive exams.

Percutaneous intervention has been the method of choice for the treatment of TRAS with satisfactory results and few short-term complications, and its efficacy has been demonstrated, especially when using stents, in the various case series published in the literature. However, there is little data on long-term intervention, showing reduced mortality and graft preservation.

Evaluated data from the 2000-2005 United States Renal Data System (USRDS) and found no differences in mortality or renal loss in patients undergoing TRAS angioplasty (145 patients) compared to those who only underwent clinical treatment (678 patients) .

In a recently published systematic review, the authors demonstrated that percutaneous intervention with or without stenting was effective in the treatment of TRAS, with favorable results in terms of technical success (over 90%), clinical success, long graft patency, with few serious complications described. However, the authors report the absence of well-designed robust randomized studies, most of which are retrospective series of a single center with a low casuistic. The positive findings of this review contrast with the results found in the treatment of native renal artery stenosis, where stent revascularization showed no benefit in patients with atherosclerotic renovascular disease when compared to drug treatment. In this same article, the authors describe the inconsistency and lack of standardization in the methodology for defining the outcomes of the intervention on TRAS.

The Hospital do Rim e Hipertensão, an agency linked to the Federal University of São Paulo (Unifesp) in Brazil, is the world leader in renal transplantation, performing an average of 1000 transplants / year in recent years. From 2006 to January 2015, patients with suspected TRAS were referred for angiography in the Hemodynamics of Hospital São Paulo.

The aims of this study was to retrospectively evaluate all patients referred to service with suspected TRAS who underwent angiography and intervention.

ELIGIBILITY:
Inclusion Criteria:

* patients with clinical suspicion of transplanted renal artery stenosis.
* patients undergoing angiography of the transplanted renal artery.
* patients undergoing transplanted renal artery stenosis intervention with and without stent.

Exclusion Criteria:

* refuses to participate in the study.
* patients without clinical follow-up.
* patients who did not renal transplanted at the hospital do Rim.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with suspected transplanted renal artery stenosis and referred to the hemodynamics laboratory for angiography of the transplanted renal artery.
Sampling Method: Non-Probability Sample
Enrollment: 313 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
overall mortality rate | 08 years
  overall mortality rate at the end of follow-up
graft failure rate | 08 years
  graft failure rate at the end of follow-up

SECONDARY OUTCOMES:
systolic and diastolic pressure measurement in mmHg | 01 month and 01 year
  systolic and diastolic pressure measurement in mmHg at 01 month and 01 year
glomerular filtration rate in mL/min/1,73 m2 | 01 month and 01 year
  glomerular rate at 01 month and 01 year in mL/min/1,73 m2

CONTACTS AND LOCATIONS:
Overall Officials: Adriano HP Barbosa, MDPhD, Study Chair — Unifesp/EPM
Locations (2):
- Brazil (2):
  - Adriano H. P. Barbosa, São Paulo, São Paulo
  - Solange Regina Generozo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Patel NH, Jindal RM, Wilkin T, Rose S, Johnson MS, Shah H, Namyslowski J, Moresco KP, Trerotola SO. Renal arterial stenosis in renal allografts: retrospective study of predisposing factors and outcome after percutaneous transluminal angioplasty. Radiology. 2001 Jun;219(3):663-7. doi: 10.1148/radiology.219.3.r01jn30663. PMID 11376251
- [Result] Henning BF, Kuchlbauer S, Boger CA, Obed A, Farkas S, Zulke C, Scherer MN, Walberer A, Banas M, Kruger B, Schlitt HJ, Banas B, Kramer BK. Percutaneous transluminal angioplasty as first-line treatment of transplant renal artery stenosis. Clin Nephrol. 2009 May;71(5):543-9. PMID 19473615
- [Result] Ngo AT, Markar SR, De Lijster MS, Duncan N, Taube D, Hamady MS. A Systematic Review of Outcomes Following Percutaneous Transluminal Angioplasty and Stenting in the Treatment of Transplant Renal Artery Stenosis. Cardiovasc Intervent Radiol. 2015 Dec;38(6):1573-88. doi: 10.1007/s00270-015-1134-z. Epub 2015 Jun 19. PMID 26088719
- [Result] Valpreda S, Messina M, Rabbia C. Stenting of transplant renal artery stenosis: outcome in a single center study. J Cardiovasc Surg (Torino). 2008 Oct;49(5):565-70. PMID 18670375
- [Result] Marini M, Fernandez-Rivera C, Cao I, Gulias D, Alonso A, Lopez-Muniz A, Gomez-Martinez P. Treatment of transplant renal artery stenosis by percutaneous transluminal angioplasty and/or stenting: study in 63 patients in a single institution. Transplant Proc. 2011 Jul-Aug;43(6):2205-7. doi: 10.1016/j.transproceed.2011.06.049. PMID 21839234
- [Result] Peregrin JH, Stribrna J, Lacha J, Skibova J. Long-term follow-up of renal transplant patients with renal artery stenosis treated by percutaneous angioplasty. Eur J Radiol. 2008 Jun;66(3):512-8. doi: 10.1016/j.ejrad.2007.05.029. Epub 2007 Jul 12. PMID 17629433
- [Result] Su CH, Lian JD, Chang HR, Wu SW, Chen SC, Tsai CF, Kao PF, Ueng KC. Long-term outcomes of patients treated with primary stenting for transplant renal artery stenosis: a 10-year case cohort study. World J Surg. 2012 Jan;36(1):222-8. doi: 10.1007/s00268-011-1312-3. PMID 22045446
- [Result] Ali A, Mishler D, Taber T, Agarwal D, Yaqub M, Mujtaba M, Goggins W, Sharfuddin A. Long-term outcomes of transplant recipients referred for angiography for suspected transplant renal artery stenosis. Clin Transplant. 2015 Sep;29(9):747-55. doi: 10.1111/ctr.12574. Epub 2015 Jul 14. PMID 26052624
- [Result] Hurst FP, Abbott KC, Neff RT, Elster EA, Falta EM, Lentine KL, Agodoa LY, Jindal RM. Incidence, predictors and outcomes of transplant renal artery stenosis after kidney transplantation: analysis of USRDS. Am J Nephrol. 2009;30(5):459-67. doi: 10.1159/000242431. Epub 2009 Sep 24. PMID 19776559
- [Result] Sharma S, Potdar A, Kulkarni A. Percutaneous transluminal renal stenting for transplant renal artery stenosis. Catheter Cardiovasc Interv. 2011 Feb 1;77(2):287-93. doi: 10.1002/ccd.22758. PMID 20824760
- [Result] Willicombe M, Sandhu B, Brookes P, Gedroyc W, Hakim N, Hamady M, Hill P, McLean AG, Moser S, Papalois V, Tait P, Wilcock M, Taube D. Postanastomotic transplant renal artery stenosis: association with de novo class II donor-specific antibodies. Am J Transplant. 2014 Jan;14(1):133-43. doi: 10.1111/ajt.12531. PMID 24354873
- [Result] Audard V, Matignon M, Hemery F, Snanoudj R, Desgranges P, Anglade MC, Kobeiter H, Durrbach A, Charpentier B, Lang P, Grimbert P. Risk factors and long-term outcome of transplant renal artery stenosis in adult recipients after treatment by percutaneous transluminal angioplasty. Am J Transplant. 2006 Jan;6(1):95-9. doi: 10.1111/j.1600-6143.2005.01136.x. PMID 16433762
- [Result] Seratnahaei A, Shah A, Bodiwala K, Mukherjee D. Management of transplant renal artery stenosis. Angiology. 2011 Apr;62(3):219-24. doi: 10.1177/0003319710377076. Epub 2010 Aug 3. PMID 20682611
- [Result] Voiculescu A, Schmitz M, Hollenbeck M, Braasch S, Luther B, Sandmann W, Jung G, Modder U, Grabensee B. Management of arterial stenosis affecting kidney graft perfusion: a single-centre study in 53 patients. Am J Transplant. 2005 Jul;5(7):1731-8. doi: 10.1111/j.1600-6143.2005.00927.x. PMID 15943633
- [Result] Ghirardo G, De Franceschi M, Vidal E, Vidoni A, Ramondo G, Benetti E, Motta R, Ferraro A, Zanon GF, Miotto D, Murer L. Transplant renal artery stenosis in children: risk factors and outcome after endovascular treatment. Pediatr Nephrol. 2014 Mar;29(3):461-7. doi: 10.1007/s00467-013-2681-7. Epub 2013 Dec 5. PMID 24305958
- [Result] Bruno S, Remuzzi G, Ruggenenti P. Transplant renal artery stenosis. J Am Soc Nephrol. 2004 Jan;15(1):134-41. doi: 10.1097/01.asn.0000099379.61001.f8. PMID 14694165
- [Derived] Faccinetto ACB, Santos GRF, Taguchi JC, Orellana HC, Galhardo A, Kanhouche G, Barteczko MLM, Tedesco Junior H, Bravo-Valenzuela NJM, Moises VA, Pestana JOM, Silva CMC, Barbosa AHP. Retrospective analysis of percutaneous intervention of the renal artery in transplanted kidneys in children and adolescents at a tertiary public hospital. PLoS One. 2024 Mar 29;19(3):e0297975. doi: 10.1371/journal.pone.0297975. eCollection 2024. PMID 38551934
- [Derived] Kanhouche G, Santos GRF, Orellana HC, Galhardo A, Faccinetto ACB, Barteczko MLM, de Carvalho LSF, Taddeo JB, Foresto RD, Moises VA, Tedesco-Silva H, Pestana JM, Barbosa AHP. Risk factors of transplant renal artery stenosis in kidney transplant recipients. Clinics (Sao Paulo). 2022 Aug 2;77:100087. doi: 10.1016/j.clinsp.2022.100087. eCollection 2022. PMID 35931001